CLINICAL TRIAL: NCT02011334
Title: A MULTICENTER, OPEN LABEL STUDY TO EVALUATE EFFICACY AND SAFETY OF TOCILIZUMAB GIVEN SUBCUTANEOUSLY IN MONOTHERAPY AND IN COMBINATION WITH NON-BIOLOGIC DMARDS IN PATIENTS WITH MODERATE TO SEVERE ACTIVE RHEUMATOID ARTHRITIS IN LATIN AMERICA
Brief Title: A Study Assessing the Safety and Efficacy of Subcutaneous RoActemra/Actemra Alone or in Combination With Non-biologic Antirheumatics in Rhuematoid Arthritis Patients in Latin America With Inadequate Response to Non-biologic Antirheumatic Drugs.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28700
Record Dates: First submitted 2013-12-04; First posted 2013-12-13 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- RoActemra/Actemra (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 162 mg will be administered once weekly by subcutaneous injection.

SUMMARY:
This multi-center, open-label, single-arm, Phase IIIb study will evaluate the safety and efficacy of subcutaneous RoActemra/Actemra alone or in combination with non-biologic disease modifying antirheumatic drugs (DMARDs) in rheumatoid arthritis patients in Latin America with an inadequate response to non-biologic DMARDs.

ELIGIBILITY:
Inclusion Criteria:

* Patients >/= 18 years of age.
* Patients with a diagnosis of active RA according to the revised (1987) ACR criteria or EULAR/ACR (2010) criteria.
* Patients with moderate to severe RA (DAS-ESR 28 >/= 3.2).
* Receiving non-study treatment on an outpatient basis.
* Oral corticosteroids (</= 10 mg/day prednisone or equivalent), NSAIDs and non-biologic DMARDs are permitted if on a stable dose regimen for >/= 4 weeks prior to Baseline.
* Inadequate response to previous non-biologic DMARD therapy.
* Use of effective contraception throughout the study as defined by protocol; female patients of childbearing potential cannot be pregnant.

Exclusion Criteria:

* Presence of clinically significant medical conditions.
* History of diverticulitis, diverticulosis requiring antibiotic treatment, or chronic ulcerative lower GI disease that might predispose to perforation.
* Current or history of recurrent bacterial, viral, fungal, mycobacterial, or other infections.
* Any infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of Screening or oral antibiotics within 2 weeks of Screening.
* Clinically significant findings on lab tests and/or hepatits B or C, or HIV screenings.
* Active TB requiring treatment within the previous 3 years.
* Evidence of active malignant disease, malignancies diagnosed within the previous 10 years, or breast cancer diagnosed within the previous 20 years.
* History of alcohol, drug, or chemical abuse within 1 year prior to Screening.
* Neuropathies or other conditions that might interfere with pain evaluation.
* Major surgery (including joint surgery) within 8 weeks prior to Screening or planned major surgery within 6 months following Baseline.
* Rheumatic autoimmune disease other than RA, including systemic lupus erythematosis, mixed connective tissue disorder, scleroderma, polymyositis, or significant systemic involvement secondary to RA (e.g., vasculitis, pulmonary fibrosis or Felty's syndrome). Secondary Sjögren's syndrome with RA is permitted.
* Functional Class IV as defined by the ACR Classification of Functional Status in-Rheumatoid Arthritis (Appendix 2).
* Diagnosis of juvenile idiopathic arthritis or juvenile RA, and/or RA before the age of 16.
* Prior history of or current inflammatory joint disease other than RA.
* Previous exposure to RoActemra/Actemra (either IV or SC).
* Prior treatment with a biologic agent.
* Treatment with any investigational agent within 4 weeks (or five half-lives of the investigational drug, whichever is longer) of Screening.
* Previous treatment with any cell-depleting therapies, including investigational agents or approved therapies, with alkylating agents such as chlorambucil, or with total lymphoid irradiation.
* Treatment with IV gamma globulin, plasmapheresis within 6 months of Baseline.
* Immunization with a live/attenuated vaccine within 4 weeks prior to Baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2014-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Efficacy: Disease Activity Score 28-erythrocyte sedimentation rate (DAS28-ESR) Remission Rate | 24 weeks

SECONDARY OUTCOMES:
Safety: Incidence of adverse events (AE) | 60 weeks
Efficacy: Change in DAS28-ESR | From baseline to Week 52
Efficacy: ACR/EULAR responses | 52 weeks
Efficacy: Change in disease activity (CDAI/SDAI) | From baseline to Week 52
Efficacy: Change in joint swelling/tenderness (SJC/TJC) | From baseline to Week 52
Safety: Assessment of immunogenicity | 60 weeks
Patient-reported outcomes | 60 weeks
Efficacy: DAS28-ESR Remission Rate | 52 weeks
Efficacy: Proportion of patients who maintain DAS28 Remission/LDA | From Week 24 to Week 52
Safety: Rates of AE leading to dose modification or study withdrawal | 52 weeks
Safety: Assessment of physical examination and vital signs | 52 weeks
Safety: Incidence of clinically significant laboratory abnormalities following treatment | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- Argentina (4):
  - Buenos Aires
  - C. A. B. A.
  - Córdoba
  - Rosario
- Brazil (6):
  - Goiânia, Goiás
  - Cuiabá, Mato Grosso
  - Juiz de Fora, Minas Gerais
  - Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
- Colombia (3):
  - Bogota D.C.
  - Bucaramanga
  - Medellín
- Santo Domingo, Dominican Republic
- Mexico (3):
  - Mexico City
  - Mérida
  - Morelia
- Venezuela (2):
  - Maracaibo
  - Punto Fijo

REFERENCES:
- [Derived] Mysler E, Cardiel MH, Xavier RM, Lopez A, Ramos-Esquivel A. Subcutaneous Tocilizumab in Monotherapy or in Combination With Nonbiologic Disease-Modifying Antirheumatic Drugs in Latin American Patients With Moderate to Severe Active Rheumatoid Arthritis: A Multicenter, Phase IIIb Study. J Clin Rheumatol. 2020 Oct;26(7S Suppl 2):S180-S186. doi: 10.1097/RHU.0000000000001361. PMID 32251060
- [Derived] Choy E, Caporali R, Xavier R, Fautrel B, Sanmarti R, Bao M, Devenport J, Petho-Schramm A. Effects of concomitant glucocorticoids in TOZURA, a common-framework study programme of subcutaneous tocilizumab in rheumatoid arthritis. Rheumatology (Oxford). 2019 Jun 1;58(6):1056-1064. doi: 10.1093/rheumatology/key393. PMID 30649524
- [Derived] Choy E, Caporali R, Xavier R, Fautrel B, Sanmarti R, Bao M, Bernasconi C, Petho-Schramm A. Subcutaneous tocilizumab in rheumatoid arthritis: findings from the common-framework phase 4 study programme TOZURA conducted in 22 countries. Rheumatology (Oxford). 2018 Mar 1;57(3):499-507. doi: 10.1093/rheumatology/kex443. PMID 29244149